CLINICAL TRIAL: NCT04085068
Title: Effect of Dural Release on Women With Back and Neck Pain After Obstetrics and Gynecological Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, assistant lectrure, Cairo University
Other Study IDs: P.T.REC/012/00191
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group (group A):: 15 women take cranioscaral treatment
  Interventions: Other: cranioscaral treatment
- control group (group B):: shame group

INTERVENTIONS:
Other: cranioscaral treatment — dural release
  Groups: Study group (group A):

SUMMARY:
Something must be done in order to release the tension within the dura mater before any lasting correction of the spine can be effected. Each of the cranial nerves is wrapped in a sheath of dura mater. As they exit the cranial vault they are described by Gray's Anatomy as having a "dural cuff".

ELIGIBILITY:
Inclusion Criteria:

* The age of the participants will be ranged from 20 to 40 years. Their body mass index will be ranged from 20 to 25 kg/m2. They will have regular menstrual cycle. They will not receive any hormonal therapy or taking any regular drugs.

Exclusion Criteria:

* Bone disease. Discogenic state with radiculopathy or not. Systemic disease of musculoskeletal system. Any sensory problems. Previous vertebral fractures. Major spinal structural abnormality.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 30 women will participate in this study, thirty women diagnosed as having back ar neck pain after surgery.They will be selected from outpatient clinic of obstetrics and Gynaecology department in El-Hosary family health Centre.
  All participants will be given a full explanation of the protocol of the study and informed consent form will be signed from each subject before participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-11 (Estimated)

PRIMARY OUTCOMES:
body mass index | 3 months
  BMI in kg/m^2
Satisfaction assessed by the VAS | 3 months
  Degrees of menstrual pain will be assessed using a VAS, which was a method of representing subjects' pain on a 10 cm linear scale. Score of 0 meant 'no pain' and 10 meant 'worst pain'. Tomeasure specific symptoms
a pressure-pain threshold | 3 months
  algometer Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. It has been noted in pressure-pain threshold studies that the rate at which manual force is applied should be consistent to provide the greatest reliability

IPD SHARING:
Plan to Share IPD: Undecided